CLINICAL TRIAL: NCT02910726
Title: Non-inferiority Study of Intra-operative Indocyanine Green Fluorescent Dye Versus Technetium Lymphoscintigraphy for Sentinel Lymph Node Biopsy in Pediatric Malignancies
Brief Title: A Study Comparing Green Fluorescent Dye and Radioactive Dye for Sentinel Lymph Node Biopsy in Pediatric Cancers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-1003
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Patients With Solid Tumors
Keywords: indocyanine green fluorescent dye; Technetium lymphoscintigraphy; sentinel lymph node biopsy; 16-1003
MeSH Terms: interventions — Sentinel Lymph Node Biopsy; Indocyanine Green

ARMS (1):
- Sentinel Lymph Node Biopsy (Experimental): This is a single-center clinical trial to evaluate non-inferiority of ICG-guided SLN biopsy compared with the gold standard TcL-guided SLN biopsy in pediatric patients with solid tumors. Each patient will undergo TcL, consistent with the standard of care, but the surgeon will be blinded to the results preoperatively. Intraoperatively, ICG injection and transdermal lymphography will be used to identify the draining nodal basin and the position of the sentinel nodes. ICG transdermal lymphography will be considered successful if SLNs can be visualized on near-infrared imaging. After the transdermal lymphography results have been recorded, the surgeon will be unblinded to the TcL mapping.
  Interventions: Procedure: Sentinel Lymph Node Biopsy; Drug: indocyanine green (ICG)

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy
Drug: indocyanine green (ICG)

SUMMARY:
This study is being done in patients that have tumors to find out how well sentinel lymph nodes (SLNs) can be found with a special dye called indocyanine green (ICG).

ELIGIBILITY:
Inclusion Criteria:

* Patients <30 years old with an extracoelomic solid tumor, diagnosis confirmed at the enrolling institution, requiring SLN biopsy
* Women of childbearing potential must have a negative pregnancy test (urine or blood) pre-operatively as per the standard hospital policy. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant.
* Patients who are cleared for surgery

Exclusion Criteria:

* History of reaction to ICG, iodides, or technetium radiocolloid
* Intracoelomic primary tumors or tumors expected to drain to an intracoelomic SLN
* Patients with extensive prior surgery at the primary site or nodal basin expected to affect the lymphatic drainage
* Patients unwilling or unable to sign informed consent
* Women who are pregnant or breast-feeding

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Heaton, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - St. Jude's Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Sentinel Lymph Node Biopsy: This is a single-center clinical trial to evaluate non-inferiority of ICG-guided SLN biopsy compared with the gold standard TcL-guided SLN biopsy in pediatric patients with solid tumors. Each patient will undergo TcL, consistent with the standard of care, but the surgeon will be blinded to the results preoperatively. Intraoperatively, ICG injection and transdermal lymphography will be used to identify the draining nodal basin and the position of the sentinel nodes. ICG transdermal lymphography will be considered successful if SLNs can be visualized on near-infrared imaging. After the transdermal lymphography results have been recorded, the surgeon will be unblinded to the TcL mapping.
  Sentinel Lymph Node Biopsy
  indocyanine green (ICG)
Period: Overall Study
Arm/Group | Sentinel Lymph Node Biopsy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sentinel Lymph Node Biopsy
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 15 [8 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: % of Patients in Whom a Sentinel Lymph Node is Identified
Description: These percentages will be compared using a non-inferiority comparison for matched pair data.
Time Frame: 1 year
Population: N/A - data were not collected
Arm/Group | Sentinel Lymph Node Biopsy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Sentinel Lymph Node Biopsy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/26/NCT02910726/Prot_SAP_000.pdf